CLINICAL TRIAL: NCT06716749
Title: Effectiveness of Adding Morphine to Intraosseous Vancomycin for Pain Control in Total Knee Arthroplasty: A Double-Blind, Randomized Trial
Brief Title: Effectiveness of Adding Morphine to Intraosseous Vancomycin for Pain Control in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB-24-1831
Record Dates: First submitted 2024-11-17; First posted 2024-12-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Primary Total Knee Arthroplasty; Intraosseous Morphine Injection; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Morphine; Vancomycin

STUDY DESIGN:
Intervention Model Description: 43 patients receiving placebo. 43 patients receiving experimental.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, care team, and research team are all blinded to their respective group until the study is concluded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Intraosseous vancomycin with no morphine) (Placebo Comparator): Control patients will receive 500 mg of vancomycin in 100 mL of normal saline + 10 mL of normal saline (placebo). Both with be injected intraosseously in the tibia.
  Interventions: Drug: Vancomycin
- Experimental (Intraosseous vancomycin with morphine) (Experimental): Control patients will receive 500 mg of vancomycin in 100 mL of normal saline + 10 mg of morphine in 10 mL of normal saline. Both with be injected intraosseously in the tibia.
  Interventions: Drug: Morphine; Drug: Vancomycin

INTERVENTIONS:
Drug: Morphine — 10 mg morphine in 10 mL normal saline
  Other Names: IO pain medication
  Arms: Experimental (Intraosseous vancomycin with morphine)
Drug: Vancomycin — 500 mg Vancomycin in 100 mL of normal saline
  Other Names: IO antibiotic

SUMMARY:
Study investigators propose to investigate if a bony injection of pain medication during a knee replacement will help pain levels following primary knee replacement surgery. To investigate this, 86 patients will be enrolled. Half of the patients will receive a bony injection of antibiotics with morphine (pain medication) while the other half will receive a bony injection of antibiotics with placebo (no pain medication). Following surgery, patient pain levels and pain medication consumption will be measured.

The injection is intraosseous meaning in the bone. The needle pierces the bone and the medication is injected into the bone. The site of injection is on the anterior (front) of the upper portion of the tibia. The medications are Vancomycin (antibiotic) and Morphine (pain medication) which are mixed in separate syringes and then injected. Intraosseous vancomycin is standard of care while intraosseous vancomycin with morphine is also standard of care, depending on operating surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. 18-100 years old
2. Primary total knee arthroplasty
3. Participants must be able to consent for themselves
4. Capable and comfortable with text messaging

Exclusion Criteria:

1. Non-primary total knee arthroplasty
2. Intraoperative or postoperative deviation from standard of care
3. Post-traumatic surgical indication
4. Post-infectious surgical indication
5. Chronic narcotic use or history of narcotic addiction
6. Allergy to vancomycin
7. Allergy to morphine
8. Inability to receive spinal anesthesia
9. Inability to receive intraoperative adductor canal block
10. Inability to provide informed consent for the study
11. Inability to speak English fluently

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Postoperative pain levels | 14 days postoperatively
  Pain scores on a scale of 0-10 with 0 meaning no pain and 10 being the worst pain possible
Postoperative pain medication consumption | 14 days postoperatively
  How much pain medication patients consumed following surgery. Measured in morphine milliequivalents (MME).

SECONDARY OUTCOMES:
Number of patients with postoperative nausea and vomiting | 14 days postoperatively
  Number of patients with postoperative nausea and vomiting episodes within 14 days of surgery
Patient reported outcomes (KOOS) | 1 month preoperative to 6 weeks postoperative
  Patient reported outcomes preoperative and postoperative. Preoperative measurement compared to 6 weeks postoperative. KOOS is measured 0-100 with 0 representing total knee disability and 100 representing a perfect knee.
Patient reported outcomes (PROMIS) | 1 month preoperative to 6 weeks postoperative
  Patient reported outcomes preoperative and postoperative. Preoperative measurement compared to 6 weeks postoperative.
  Range is 20-80 with higher being better. The mean is 50 with the standard deviation being 10.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph T Moskal, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States